CLINICAL TRIAL: NCT04604951
Title: Below the Belt: Non-invasive Neuromodulation to Treat Bladder, Bowel, and Sexual Dysfunction Following Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: International Spinal Research Trust (Other); International Collaboration on Repair Discoveries (Other); Providence Health & Services (Other)
Responsible Party: Principal Investigator, Andrei Krassioukov, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H20-01163; 2019-1092 (Other Grant/Funding Number: International Spinal Research Trust)
Record Dates: First submitted 2020-09-28; First posted 2020-10-27 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Spinal Cord Injuries; Neurogenic Bladder; Neurogenic Bowel; Spinal Cord Stimulation; Sexual Dysfunction, Physiological
Keywords: Transcutaneous Spinal Cord Stimulation; Noninvasive Spinal Cord Stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic; Neurogenic Bowel; Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate (Experimental): Group 1: Moderate 2 times per week transcutaneous spinal cord stimulation.
  Interventions: Device: Transcutaneous Spinal Cord Stimulation
- Intensive (Experimental): Group 2: Intensive 5 times per week transcutaneous spinal cord stimulation.
  Interventions: Device: Transcutaneous Spinal Cord Stimulation

INTERVENTIONS:
Device: Transcutaneous Spinal Cord Stimulation — This non-invasive therapeutic modality uses electrodes applied over the skin to deliver electrical stimulation. It is based on the same principles of ground-breaking work from the investigator's group and others, showing that stimulation of the spinal cord can promote motor and autonomic (cardiovascular, bladder, bowel) recovery in individuals with chronic SCI.
  Other Names: Noninvasive spinal cord stimulation

SUMMARY:
Recent findings have demonstrated that electrical stimulation to the spinal cord (i.e. implanted electrodes) can significantly recover bladder, bowel, and sexual function after injury. While promising, a major drawback is that individuals must undergo a highly invasive and expensive surgical procedure to implant the stimulator on top of the spinal cord. Moreover, the inability to re-position the implanted stimulator considerably limits the flexibility of this procedure.

In this project, the investigators propose a comprehensive clinical study examining the effects of TCSCS in promoting recovery of these crucial functions in individuals with spinal cord injury (SCI). This non-invasive therapeutic modality uses electrodes applied over the skin to deliver electrical stimulation. It is based on the same principles of ground-breaking work from the investigator's group and others, showing that stimulation of the spinal cord can promote motor and autonomic (cardiovascular, bladder, bowel) recovery in individuals with chronic SCI.

DETAILED DESCRIPTION:
For decades, clinicians and scientists have focused on finding a cure for paralysis. However, research has shown that individuals with SCI more highly prioritize bladder, bowel and sexual functioning over the ability to walk again. There is still a major lack of research towards improving these critical components of autonomic recovery following SCI. This clinical study examines the EFFECTS OF TRANSCUTANEOUS SPINAL CORD STIMULATION (TCSCS) in promoting recovery of bladder, bowel and sexual functions in individuals with SCI. This NON-INVASIVE THERAPEUTIC METHOD utilizes electrodes applied over the skin, and is based on ground-breaking work (from the investigator's group and others), showing that spinal cord stimulation can promote motor and autonomic recovery in individuals with chronic SCI. This study is a collaborative effort between clinicians and scientists with expertise in: SCI care, rehabilitation, bladder, bowel, cardiovascular and sexual functioning.

Safety will be routinely monitored. Six weeks after completion of stimulation experiments, bladder, bowel and sexual function will be reassessed to examine the longevity of TCSCS-induced effects. TCSCS COULD OFFER A SIMPLE, COST-EFFECTIVE SOLUTION TO TREAT AUTONOMIC DYSFUNCTIONS (i.e. urine and faecal incontinence, erectile difficulties etc.) that would undoubtedly significantly improve overall health related quality of life for individuals with SCI.

Recent findings have demonstrated that electrical stimulation to the spinal cord (i.e. implanted electrodes) can significantly recover bladder, bowel, and sexual function after injury. While promising, a major drawback is that individuals must undergo a highly invasive and expensive surgical procedure to implant the stimulator on top of the spinal cord. Moreover, the inability to re-position the implanted stimulator considerably limits the flexibility of this procedure.

In this project, the investigators propose a comprehensive clinical study examining the effects of TCSCS in promoting recovery of these crucial functions in individuals with SCI. This non-invasive therapeutic modality uses electrodes applied over the skin to deliver electrical stimulation. It is based on the same principles of ground-breaking work from the investigator's group and others, showing that stimulation of the spinal cord can promote motor and autonomic (cardiovascular, bladder, bowel) recovery in individuals with chronic SCI.

Electrical neuromodulation has recently emerged as a leader in potential therapies for restoring voluntary control of functional movements in lower limbs after SCI. In addition to functional motor recovery, numerous studies from the investigator's group and collaborators have shown efficacy of both epidural stimulation (invasive) and non-invasive stimulation (TCSCS) in restoring autonomic function. For example, in the investigators preliminary examination of several individuals with SCI, the investigators have demonstrated that epidural stimulation acutely restores cardiovascular control, improves lower urinary tract (LUT) function and reduces time needed for bowel routine. These studies were highly influential in developing stimulation protocols and establishing spinal cord stimulation as a safe and effective therapy. The next logical step is to conduct a wider-scale clinical trial for TCSCS as a novel, efficacious and inexpensive alternative therapy to epidural stimulation. By uniting experts in the field of SCI, physical medicine/rehabilitation, urology, colorectal health and sexual functioning, the investigators are well-equipped to assess TCSCS as a novel means of improving recovery of LUT, bowel and sexual function. The investigator's team has a strong history of collaborative research in these fields and extensive experience in the evaluation of these three aspects of autonomic function using physiological measures/clinical assessments in addition to well-validated questionnaires.

The investigators anticipate that individuals with SCI who participate in this trial will receive a therapeutic benefit in at least one of the multiple outcomes (i.e. LUT, bowel and sexual function) and will also obtain greater insight into the nature of their current health status in these areas post-SCI. This project will also have a high degree of impact on the SCI-community by further developing TCSCS as a more accessible and inexpensive therapy for autonomic dysfunctions. Ultimately the investigator's goal is to improve quality of life for individuals with SCI, which the investigators anticipate in turn will decrease caregiver burden and health care costs due to LUT, bowel and sexual issues associated with SCI.

Eligible individuals who sign the consent form will first undergo screening and initial evaluations (total of 6 visits completed within 6 weeks) and then will be randomly assigned to either a moderate TCSCS treatment group (2 days/week for a total of 12 treatment sessions) or intense TCSCS treatment group (5days/week for a total of 30 treatment sessions) during the 6 weeks treatment period. After completion of total protocol, each participant will undergo 4 follow up assessments that will be completed within 12 weeks following the treatment. Overall, the total duration of participation will be approximately 25 weeks.

Visit 1 Screening Approximately 1.5 hours After a participant has provided informed consent, he/she will be assigned a unique study number will be invited for a screening assessment to confirm study eligibility.

Visit 2: Baseline Assessments Approximately 1 hour. All eligible participants will be guided through a series of questionnaires on bladder function, bowel function, cardiovascular function and sexual health (outcomes 6-10 below). Participants will also undergo baseline 24 hours ambulatory evaluation of cardiovascular functions (outcome 1).

Visit 3 /Baseline EMG Mapping of Spinal Cord Segments with TCSCS Approximately 2 hours. Participants will undergo baseline mapping using surface EMG and concentric needle EMG as per an established protocol to record muscle activation during transcutaneous spinal cord stimulation (mapping) at different spinal cord levels and different intensity (outcome 2).

Visits 4,5 and 6: Bladder and bowel function assessment procedures with and without non-invasive transcutaneous spinal cord stimulation Approximately 2.5 hours per visit.

Visits 4, 5, and 6 will include assessments of bladder function (urodynamics, outcome 3) and bowel function (Anorectal Manometry, outcome 4). Bladder assessments will take place at the Blusson Spinal Cord Centre and bowel assessments will take place at St. Paul's Hospital.

The order of these 3 visits will differ randomly between individuals and will be one of the following:

* Pathway #1: you will start with Urodynamics, (UDS 1, Visit 4), followed by a second session of Urodynamics (UDS 2, Visit 5), followed by bowel function assessments(Visit 6).
* Pathway#2: you will start bowel function assessments (Visit 4), followed by Urodynamics (UDS 1, Visit 5), and a second session of Urodynamics (UDS 2, Visit 6)).

Visits 7-18 or 36: Long Term Non-invasive transcutaneous spinal cord stimulation Approximately 1.5 hours per visit.

Participants will be asked to come to ICORD for TCSCS either 2 days/week (moderate treatment group with total 12 treatment sessions) or 5 days/week (intense treatment group with total 30 treatment sessions) for 6 weeks. Participants will be randomly assignment to either the moderate or intense treatment groups. Whether a participant are assigned to the moderate or intense group will be determined by chance (like the flip of a coin). Each TCSCS session will last approximately 90 minutes. Stimulation will be applied for a total of 60 minutes in three 20-minute intervals with 2 minute breaks. Skin temperature, blood pressure and heart rate will be monitored. Mid-way through the 6 weeks, participants will be set up with an ambulatory blood pressure monitor to wear at home on the day of the participant's bowel routine. We will also provide a diary for participants to log their activities while wearing the blood pressure monitor.

Visit 19 or 37: Bladder assessment and SCI severity assessment - Approximately 3 hours

After the 6 weeks of TCSCS, a third urodynamics assessment will be performed at the Blusson Spinal cord centre, following the same procedure described above, both without and with TCSCS. During this visit, a clinician will also perform a SCI severity assessment (International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) exam).

Visit 20 or 38: Immediate Follow up Telephone Questionnaires - Approximately 1 hour

Visit 20 or 38 will take place by telephone or video conference call (considering the present COVID-19 pandemic environment). Participants will be guided through the same series of questionnaires as in visit 1 and 2, on bladder function, bowel function, cardiovascular function and sexual health.

Visits 21-22 or 39-40: Long Term follow up Telephone Questionnaires and Semi Structured Interview:

Approximately 1 hour (visit 21/39) and approximately 1.5 hours (visit 22/40)

These visits will take place over the telephone to evaluate existing and new adverse events and concurrent treatments. During each of these follow-up phone Visits (39 and 40) at 6 and 12 weeks post completion of long term TCSCS, participants will be guided through the same series of questionnaires on bladder function, bowel function, cardiovascular function and sexual health described above.

During visit 22 or visit 40, a sexual health clinician, with experience providing clinical care to individuals with SCI, will also conduct a semi-structured qualitative interview (outcome 11) during which they will ask participants questions about the following: sexual history and current relationship status, level of sexual drive, ability to orgasm, barriers to sexual activity, self-esteem, the use of performance enhancing aids, and the participant's perceptions of the role of TCSCS on sexual functioning.

ELIGIBILITY:
A participant must meet all of the following criteria in order to be eligible for inclusion:

1. Resident of British Columbia, Canada with active provincial medical services plan
2. Male or female, 18-65 years of age
3. Chronic traumatic SCI (non-progressive, with complete motor paralysis) at or above the T6 spinal segment.
4. >1-year post injury, at least 6 months from any spinal surgery.
5. Documented presence of bladder dysfunction (NDO during UDS)
6. Documented presence of bowel or sexual dysfunction.
7. American Spinal Injury Association Impairment Scale (AIS) A, B.
8. Greater than or equal to antigravity strength in deltoids and biceps bilaterally
9. Hand function sufficient to perform Clean Intermittent Catheterization (CIC) or a committed caregiver to provide CIC for management of urinary bladder drainage.
10. Participants must have documented three days of bladder and bowel history prior to their baseline visit.
11. Willing and able to comply with all clinic visits and study-related procedures. Able to understand and complete study-related questionnaires (must be able to understand and speak English or have access to an appropriate interpreter as judged by the investigator).
12. No painful musculoskeletal dysfunction, unhealed fracture, pressure sore, or active infection that may interfere with testing activities.
13. Stable management of spinal cord related clinical issues (i.e., spasticity management).
14. Women of childbearing potential must not be intending to become pregnant, currently pregnant, or lactating. The following conditions apply:
15. Women of childbearing potential must have a confirmed negative pregnancy test prior to the baseline visit. During the trial, all women of childbearing potential will undergo urine pregnancy tests at their monthly clinic visits as outlined in the schedule of events.

    Women of childbearing potential must agree to use adequate contraception*~2~* during the period of the trial and for at least 28 days after completion of treatment.
16. Effective contraception includes abstinence. Sexually active males with female partners of childbearing potential must agree to use effective contraception during the period of the trial and for at least 28 days after completion of treatment.
17. Must provide informed consent.

Exclusion Criteria:

A participant who meets any of the following criteria will be ineligible to participate:

1. Presence of severe acute medical issue that in the investigator's judgement would adversely affect the participant's participation in the study. Examples include, but are not limited to clinically significant renal or hepatic disease; acute urinary tract infections; pressure sores; active heterotopic ossification; newly changed antidepressant medications [tricyclics]; or unstable diabetes. The following conditions apply:

   1. Moderate and severe forms of renal dysfunctions (eGFR below 60 ml/min)
   2. Clinically significant abnormal laboratory tests (ALT; Alkaline Phosphatase; Bilirubin [total]; GGT) as judged by the investigator.
2. Recent treatment with OnabotulinumtoxinA into the detrusor muscle (within 9 months of the baseline visit)
3. Ventilator dependent
4. Clinically significant depression or ongoing drug abuse
5. Use of any medication or treatment that in the opinion of the investigator indicates that it is not in the best interest of the participant to participate in this study.
6. Intrathecal baclofen pump.
7. Cardiovascular, respiratory, bladder, or renal disease unrelated to SCI or presence of hydronephrosis or presence of obstructive renal stones.
8. Any implanted metal in trunk or spinal cord under the sites of application of electrodes (between anode and cathode) for those who are allocated to receive TCSCS.
9. Severe anemia (Hgb<8 g/dl) or hypovolemia
10. Participant is a member of the investigational team or his /her immediate family.
11. Participant has undergone electrode implantation surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Change in bladder capacity measured by urodynamics | Weeks 4-6, Week 19
  Changes from baseline during TCSCS (%) in bladder capacity will be calculated. Urodynamics will be performed with and without TCSCS during 3 separate sessions to assess the changes from baseline in the parameters listed above. These measures will be compared to assess reproducibility of changes within urodynamic parameters during TCSCS and after long-term TCSCS.
Change in resting anorectal pressure determined via anorectal manometry | Weeks 4-6
  Anorectal manometry will be performed without and with TCSCS to assess the impact of TCSCS on anorectal pressure.

SECONDARY OUTCOMES:
Surface EMG recording with TCSCS | Weeks 3-4
  EMG measurements will allow the investigators to identify the motor threshold for skeletal muscles innervated by spinal segments known to be responsive for lower urinary tract and bowel control by delivering TCSCS at various spinal cord segments: T10/T11; T11/T12; T12/L1; L1/L2 (conus medullaris), thereby generating individualized spatiotemporal activation maps.
Change in International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) score | Week 1, Week 19
  The ISNCSCI examination will be performed by an experienced and trained investigator before and after long-term TCSCS to identify change in motor and sensory impairment and severity.
Change in Autonomic Dysfunction following Spinal Cord Injury (ADFSCI) score | Week 1, Week 19
  The ADFSCI questionnaire will be used before and after the long-term TCSCS to assess change in the degree of general autonomic dysfunction.
Change in Neurogenic Bladder Symptom Score (NBSS) | Weeks 3-4, Week 19, Week 25
  The assessment of neurogenic bladder symptoms will be performed to assess the impact of long term TCSCS on this measure. Total and domain scores (incontinence, storage and voiding, and consequences) will be calculated, with higher scores representing worse symptoms.
Change in the Incontinence Quality of Life (I-QoL) score | Weeks 3-4, Week 19, Week 25
  Assessment of urinary incontinence will be performed to assess the impact of long term TCSCS on this measure. The scale is a 100 point scale where 0 is most severe incontinence.
Change in Time Needed for Bowel Movement (TNFBM) | Weeks 3-4, Week 19, Week 25
  Pre- and post-intervention bowel management times will be compared to determine the long-term effect of TCSCS on bowel function. Difference in bowel management times will be calculated.
Change in Neurogenic Bowel Dysfunction Score (NBDS) | Weeks 3-4, Week 19, Week 25
  Assessment neurogenic bowel symptoms will be performed to assess the impact of long term TCSCS on this measure. Total score will be calculated (ranging from 0 to 47), with higher scores representing worse symptoms.
Change in the modified Wexner fecal incontinence score | Weeks 3-4, Week 19, Week 25
  Assessment of fecal incontinence will be performed to assess the impact of long term TCSCS on this measure. Total score will be calculated (ranging from 0 to 20), with a higher score representing greater incontinence.
Change in the International Index of Erectile Function (IIEF) score (for male participants) | Weeks 3-4, Week 19, Week 25
  This measure of sexual function will be used to assess whether sexual function is impacted by TCSCS. Total score (ranging from 5 to 25) and domain scores (erectile function, orgasmic function, intercourse satisfaction, and overall satisfaction) will be calculated, with higher scores representing greater function.
Change in the Female Sexual Function Index (FSFI) score (for female participants) | Weeks 3-4, Week 19, Week 25
  This measure of sexual function will be used to assess whether sexual function is impacted by TCSCS. Total score (ranging from 2 to 36) and domain scores (desire, arousal, lubrication, orgasm, satisfaction, and pain) will be calculated, with higher scores representing greater function.
Change in subjective sexual function will be measured using semi-structured interview | Week 19
  A sexual health clinician, with experience providing clinical care to individuals with SCI, will conducts a semi-structured qualitative interview at trial completion to measure change in subjective sexual function and satisfaction.
Change in 24-hour blood pressure monitoring | Weeks 3-4, Week 19
  Pre- and post-intervention 24-hour blood pressure monitoring will be compared to determine the long-term effect of TCSCS on blood pressure.
Blood pressure will be measured continuously during TCSCS | Weeks 3-18
  Continuous blood pressure monitoring will be utilized as a safety measure to detect potential adverse cardiovascular events (ACVEs, e.g., autonomic dysreflexia).

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Krassioukov, MD,PhD,FRCPC, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Blusson Spinal Cord Centre, Vancouver, British Columbia
  - St Paul's Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No